CLINICAL TRIAL: NCT06729814
Title: Prospective Assessment of Acute Skin Toxicities in Breast Cancer Patients Undergoing Retreatment with 40 Gy in 15 Fractions Radiation Therapy
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Irene Karam, Radiation Oncologist, Sunnybrook Health Sciences Centre
Other Study IDs: Prospective Study
Record Dates: First submitted 2024-08-27; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Radiation Dermatitis
Keywords: Prospective; acute skin toxicities; Quality of Life
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The most common cancer affecting Canadian women is breast cancer, with an estimated 1 in 8 women expected to be diagnosed with breast cancer during their lifetime. Improved screening and treatment have decreased mortality of breast cancer patients, however 14% of cancer-related deaths in Canadian women are still due to breast cancer. Common treatments for breast cancer include surgery, chemotherapy, hormone therapy, and radiation therapy (RT).

Despite recent improvements in treatment and preventative screenings, 20% of breast cancer patients will develop local disease recurrence or another ipsilateral primary breast cancer. . The optimal treatment of recurrent or new primary breast cancers for patients who have undergone prior radiotherapy (RT) is not well-defined. Common treatment approaches consist of mastectomy or a second breast conserving surgery (BCS) with whole or partial breast reirradiation (reRT). In the past, mastectomy has been the preferred treatment for recurrent breast cancer due to concerns over serious acute and late skin toxicities that may result from additional reRT. Many of these late skin toxicities, such as fibrosis, are chronic and can result in patients experiencing pain or other negative impacts to quality of life (QOL).

DETAILED DESCRIPTION:
Despite recent improvements in treatment and preventative screenings, 20% of breast cancer patients will develop local disease recurrence or another ipsilateral primary breast cancer. The optimal treatment of recurrent or new primary breast cancers for patients who have undergone prior radiotherapy (RT) is not well-defined. Common treatment approaches consist of mastectomy or a second breast conserving surgery (BCS) with whole or partial breast reirradiation (reRT). In the past, mastectomy has been the preferred treatment for recurrent breast cancer due to concerns over serious acute and late skin toxicities that may result from additional reRT. Many of these late skin toxicities, such as fibrosis, are chronic and can result in patients experiencing pain or other negative impacts to quality of life (QOL).

Currently at our centre, the regimen for recurrent breast cancer has been whole or partial (preferred) breast irradiation with a dose fractionation of 45 Gy in 25 fractions. However, there is concern over the treatment burden and skin toxicities that this 5-week long fractionation schedule may cause. Our breast radiation group has been recently allowed to employ 40 Gy in 15 fractions as an acceptable reRT dose fractionation. Therefore, it is vital to investigate dose fractionations for breast cancer patients undergoing retreatment due to being at a high risk of developing severe RD

Furthermore, few previous studies examining breast reRT at any dose for recurrent breast cancer have collected data on patient- and clinician- reported outcomes for QOL and symptoms associated with RD. Therefore, there is a need to conduct further research on the use of hypofractionated reRT for patients with recurrent breast cancer to discover its impact on the severity of acute skin toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Informed consent
* Histological confirmation of breast malignancy (invasive or in situ carcinoma) or phyllodes
* Previous history of ipsilateral breast cancer treated with RT
* Patients are planned to receive hypofractionated (40Gy/15) RT to the whole or partial breast or chest wall
* Patients treated with or without the addition of a planned boost or bolus
* Patients receiving local or locoregional radiation treatment
* Can communicate in English or be aided by a translator

Exclusion Criteria:

* Patients scheduled to receive conventionally fractionated (50Gy/25 or 45Gy/25) or extreme hypofractionation (26Gy/5)
* Patients planned to receive brachytherapy
* Patients with active rash, pre-existing dermatitis, or other conditions within the treatment area that may make skin assessment for the study difficult per treating physician discretion
* Concomitant cytotoxic chemotherapy
* Scleroderma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent ipsilateral breast cancer who satisfy the eligibility criteria will be approached for the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-08-07 (Estimated); Study Completion 2026-08-07 (Estimated)

PRIMARY OUTCOMES:
Effects of hypofractionated reRT (40Gy in 15 fractions) on acute skin toxicity | 3 month f/u
  To examine the effects that hypofractionated reRT (40Gy in 15 fractions) has on acute skin toxicity in patients with recurrent ipsilateral breast cancer.

SECONDARY OUTCOMES:
Impact of QOL due to hypofractionated reRT for breast cancer measured via Skindex 16 | 3 month f/u
  To evaluate the development of acute skin toxicities and the impact on quality of life due to adverse events caused by using hypofractionated reRT by using the Skindex-16 assessment tool.
Impact of QOL due to hypofractionated reRT for breast cancer measured via RISRAS | 3 month f/u
  To evaluate the development of acute skin toxicities and the impact on quality of life due to adverse events caused by using hypofractionated reRT by using the RISRAS assessment tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Odette Cancer Center Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada